CLINICAL TRIAL: NCT06358612
Title: Evaluation of An Anxiety Reducing Tool During Thyroid Biopsies: A Randomized Controlled Trial
Brief Title: Evaluation of an Anxiety Reduction Tool During Thyroid Biopsies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DALNSHA2024ABR001
Record Dates: First submitted 2024-03-29; First posted 2024-04-10 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Balls (Experimental): Patients given a stress ball in each hand.
  Interventions: Other: Stress Balls
- No Stress Balls (No Intervention): Patients NOT given a stress ball in each hand.

INTERVENTIONS:
Other: Stress Balls — Patients in the experimental arm will receive a foam stress ball to squeeze during their biopsy procedure.
  Arms: Stress Balls

SUMMARY:
Patients undergoing thyroid biopsy under local anesthetic will be asked to fill out a questionnaire that evaluates their anxiety level before and after their procedure. Patients will be randomly assigned to either use an anxiety reducing tool (stress balls in each hand) to take their mind off the procedure or will not receive an anxiety reducing tool.

DETAILED DESCRIPTION:
This is a prospective, open-label randomized controlled trial. Given the nature of the intervention, it is not possible to blind participants and the health providers to the treatment group that they are randomized to. The investigators have chosen to conduct a randomized controlled trial as stress balls are not currently a standard offering during IR procedures, and implementing the intervention is relatively simple with minimal to no additional risk to participants in the treatment group. Thyroid biopsies biopsies have been selected as the procedures for this study as these are performed on a regular basis and are conducted solely under local anesthetic without the potentially confounding effect of sedation.

If stress balls are shown to be effective in reducing intraprocedural anxiety, it could become a standard offering for patients undergoing procedures exclusively under local anaesthesia. Use of this tool could also potentially reduce the need for sedation in more complex procedures. Use of a stress ball is a low-cost intervention requiring little investment if the benefit of reducing anxiety and improving patient well-being can be confirmed. Positive results may also open the door to further studies to determine its effectiveness in other anxiety-inducing procedures performed in IR.

The study will take place in the Victoria General Hospital Biopsy Room at the Diagnostic Imaging department of the QEII Health Sciences Centre in Halifax, NS. In the 2023 calendar year, 370 thyroid biopsies were performed at the Centre.

-Research Question and Hypothesis-

Research question: will patients undergoing thyroid biopsies report reduced anxiety if provided with a stress ball compared with those who do not receive one?

Hypothesis: thyroid biopsy patients who are given a stress ball during their procedure will report reduced anxiety compared with patients who do not receive one.

-Variables-

Independent variables: "stress ball" (SB) or "no stress ball" (nSB) Dependent variable: self-reported anxiety level

-Visual Analogue Scale (VAS) Questionnaires-

The VAS is a simple and easy to administer test, and has been validated for the assessment of self-perceived psychological outcomes such as pain and anxiety. The VAS consists of a continuous 100 mm horizontal rating scale, along which subjects indicate with a tick the point that they feel best represents their state at a specified time, from "not at all anxious" at 0 mm to "extremely anxious" at 100 mm. For each response, a number from 0mm - 100mm will be measured, rounded to the nearest millimeter. In this study, subjects receive a pre-procedure questionnaire and post-procedure questionnaire consisting of VAS questions among other entries. Questionnaires will also collect subject age (not specific DOB) and sex for stratified analyses.

The pre-procedure questionnaire is designed to determine baseline anxiety. It consists exclusively of VAS questions. The first question assesses the subject's current level of anxiety in anticipation of their biopsy, while the last three assess their anxiety while undergoing "routine" medical procedures.

The post-procedure questionnaire is designed to determine intraprocedural anxiety. It consists of two VAS questions: one to assess their anxiety during the procedure, and one to assess the degree to which they consider themselves an anxious person. Subjects are also offered to comment on any interventions they think could have reduced their anxiety. Questionnaires given to subjects in the SB group also has a binary yes/no question to determine whether the subject felt that the stress balls reduced their stress during the procedure.

Questionnaire pairs (pre- and post-procedure) will be pre-randomized into either the SB or nSB groups using randomization software (Random.org) and assigned a study number A-XXX (e.g., A-001). The questionnaire will directly indicate which group a participant is in. The allocation sequence will be generated by investigator NC. The radiologist will take questionnaires from the top of a stack for each subject.

-Procedure-

The radiologist performing the biopsy will ask eligible patients on arrival whether they are willing to participate in a trial investigating anxiety during biopsy procedures, and that it would entail a short questionnaire before and after the procedure where they will indicate their stress level. The patient will be informed that a non-invasive method or tool may be used during the procedure and has no harmful effects. Formal written consent will be obtained by the radiologist, at which point the subject will be enrolled in the study. All subjects will immediately fill out the pre-procedure VAS to assess their baseline anxiety level. No identifying personal health information beyond age and sex will be captured in the questionnaire.

Subjects in the SB group will receive a stress balls (in a protective plastic covering) to be held in each hand immediately prior to the procedure, and instructed to squeeze the balls whenever they feel uncomfortable or anxious. Subjects in the nSB group will not receive any intervention. Upon arrival in the recovery area, stress balls will be taken from the SB group subjects, and all participants will immediately fill out a post-procedure VAS questionnaire to assess their intraprocedural anxiety and to ask whether there are any similar interventions that they think would have improved their experience.

Overall, subjects receive the pre-procedure questionnaire immediately after they have been consented to the study. They will receive the post-procedure questionnaire upon arrival in the recovery area. The total time between each questionnaire is approximately 115 minutes, which accounts for procedure set-up, completion, and assurance that the patient is comfortable enough to leave.

-Data Collection-

Questionnaires will be collected and stored in a locked file cabinet in the Radiology Research Office (3016 Victoria Building, Victoria General Hospital). The investigator NC will collate responses and input numerical information from each response into a password-protected Excel spreadsheet housed on a password-protected USB drive to safeguard data from tampering. No personal health information other than age and sex will be recorded.

-Data Analysis-

The minimal clinically important difference (MCID) in anxiety for the study is defined as a reduction by 15% (a difference of 15mm along the 100mm VAS). This value was chosen on the basis of a study by Williams et al. (2010) that calculated this workable threshold based on the mean difference in VAS scores in patients who report a "minimal improvement" in anxiety, using the anchor-based method.

No sub-sample analyses will be conducted.

Primary Outcome Analysis

For the primary outcome, the pre-procedure VAS will collect pre-procedure anxiety (anxiety_pre), and the post-procedure VAS will collect intra-procedure anxiety (anxiety_intra). To evaluate the difference in Anxiety_intra by SB (a binary group indicator, e.g., "stress ball (SB)" vs. "non-stress ball (nSB)" patient groups) while adjusting for age, sex, Anxiety_pre, age*SB, and sex*SB, the investigators will use a multiple regression model.

A multiple linear regression model allows us to assess the effect of SB on Anxiety_intra while controlling for the other covariates (Anxiety_pre, age, sex, age*SB, and sex*SB).

Model:

Anxiety_intra = β0 + β1×SB + β2×Anxiety_pre + β3×Age + β4×Sex + β5×Sex*SB + β6×Age*SB + epsilon

* Anxiety_intra is the dependent variable.
* SB is the primary independent variable of interest (binary: SB vs. nSB).
* Anxiety_pre, age, sex, age*SB, and sex*SB are covariates.
* β0, β1, β2, β3, β4, β5, β6 are the regression coefficients.
* epsilon is the error term.

Interpreting the results:

The coefficient β1 for the variable SB will indicate the adjusted difference in Anxiety_intra between SB and nSB groups.

* If β1 is positive and statistically significant, it indicates that, on average, participants in the SB group have higher Anxiety_intra scores compared to participants in the nSB group, after adjusting for Anxiety_pre, age, sex, age*SB, and sex*SB.
* If β1 is negative and statistically significant, it suggests that participants in the SB group have lower Anxiety_intra scores compared to participants in the nSB group, holding the other variables constant.
* If β1 is not statistically significant, it implies that there is no evidence of a difference in Anxiety_intra between the SB and nSB groups after accounting for the other variables.

The coefficient β2 for the variable Anxiety_intra represents the relationship between the pre-existing anxiety levels (Anxiety_pre) and the outcome variable (Anxiety_intra), holding all other variables in the model constant. Specifically, β2 quantifies the expected change in Anxiety_intra for a one-unit increase in Anxiety_pre, after accounting for the effects of SB, age, sex, age*SB, and sex*SB.

* If β2 is positive and statistically significant, it indicates that higher pre-existing anxiety levels (Anxiety_pre) are associated with higher Anxiety_intra scores, after adjusting for the effects of SB, age, sex, age*SB, and sex*SB.
* If β2 is negative and statistically significant, it suggests that higher pre-existing anxiety levels are associated with lower Anxiety_intra scores, controlling for the other variables in the model.
* If β2 is not statistically significant, it implies that there is no evidence of a linear relationship between Anxiety_pre and Anxiety_intra, after accounting for the other variables.
* The investigators will calculate the sample mean difference and determine whether a clinically significant difference exists between the SB vs nSB groups.

Secondary Outcome Analysis

To describe (using descriptive statistics) the differences between stress ball (SB) vs no stress ball (nSB) groups in:

1. Self-perceived anxiety when undergoing other "routine" medical procedures, including dental procedures, intramuscular injections, and phlebotomy.
2. The degree to which a subject considers themselves to be an anxious person.
3. The proportion of subjects in the SB group who believe that the stress ball reduced their anxiety (assessed by a binary yes/no).
4. Age.
5. Sex.

Question 4 from the post-procedure VAS asks patients to comment on any methods they believe could have reduced their anxiety, and will be a qualitative response that will only be used to provide insights to the research team that might inform future research studies.

-Risk Management-

The investigators do not anticipate any significant complications by nature of the intervention. In the case of a previously unknown contact allergy to material in the stress ball, standard protocols for addressing the reaction will be employed.

-Knowledge Translation-

The results of the study will be disseminated by preparation of a manuscript for publication in a peer-reviewed journal. The investigators also plan to present the results at an appropriate conference or meeting to healthcare practitioners regularly involved in biopsy procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Subjects undergoing thyroid biopsies under local anesthetic that can provide consent to treatment and for the research study.

Exclusion Criteria:

1. Previous biopsy experience
2. Greater than one (1) thyroid lesion requiring biopsy
3. Known allergy or sensitivity to stress ball material or cleaning solutions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety level of greater than 15% based on Visual Analog Score (VAS) | 1 year
  The VAS is a simple and easy to administer test, and has been validated for the assessment of self-perceived psychological outcomes such as pain and anxiety. The VAS consists of a continuous 100 mm horizontal rating scale, along which subjects indicate with a tick the point that they feel best represents their state at a specified time, from "not at all anxious" at 0 mm to "extremely anxious" at 100 mm. For each response, a number from 0mm - 100mm will be measured, rounded to the nearest millimeter. In this study, subjects receive a pre-procedure questionnaire and post-procedure questionnaire consisting of VAS questions among other entries.

SECONDARY OUTCOMES:
Changes in stress ball efficacy based on anxiety during "routine" medical procedures, using VAS | 1 year
  Changes in stress ball efficacy depending on the subject's self-perceived anxiety when undergoing other "routine" medical procedures, including dental procedures, intramuscular injections, and phlebotomy.
  Measured based on individual response to VAS for each medical procedure in question (horizontal rating along 100 mm scale, ranging from 0 mm ["not at all anxious"] to 100 mm ["extremely anxious"]). Information collected here will be included in the multiple linear regression model to determine the effects of these two covariates on the primary outcome.
Changes in stress ball efficacy based on self-perceived anxiety, using VAS | 1 year
  Changes in stress ball efficacy depending on the degree to which a subject considers themselves to be an anxious person.
  Measured based on individual response to VAS asking the degree to which subject considers themselves to be an anxious person (horizontal rating along 100 mm scale, ranging from 0 mm ["not at all anxious"] to 100 mm ["extremely anxious"]). Information collected here will be included in the multiple linear regression model to determine the effects of these two covariates on the primary outcome.
Changes in stress ball efficacy based on age and sex, using questionnaire questions | 1 year
  Changes in stress ball efficacy depending on subject age and sex.
  Data collected by individual response to questionnaire. Information collected here will be included in the multiple linear regression model to determine the effects of these two covariates on the primary outcome.
Subject self-perceived change in anxiety | 1 year
  The following question will be collected and used for descriptive statistics only:
  Whether subjects will report any self-perceived change in anxiety when provided a stress ball during their procedure, regardless of the average population results (binary yes/no question). This data will be collected via questionnaire.
Subject opinion on helpful anxiety-reducing methods | 1 year
  The following question will be collected and used for descriptive statistics only:
  Survey for subjects on any methods they believe would reduce their anxiety other than the stress ball that has been provided. This data will be collected via questionnaire where the subject is given the opportunity to write out an answer.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Abraham, MD, FRCPC, Principal Investigator — Nova Scotia Health Authority/Dalhousie University
Locations (1):
- Nova Scotia Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No